CLINICAL TRIAL: NCT02894788
Title: POSTOPERATIVE INTENSIVE CARE SURVEILLANCE. A Tool to Optimize ICU-beds Management?
Brief Title: Postoperative Intensive Care Surveillance
Acronym: PoIS
Status: Completed | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: PoIS
Record Dates: First submitted 2016-07-19; First posted 2016-09-09 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Post-operative Adhesion(s)

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ICU: patients postoperatively admitted to ICU
  Interventions: Other: ICU admission
- no ICU: patients who didn't required ICU admission postoperatively

INTERVENTIONS:
Other: ICU admission
  Groups: ICU

SUMMARY:
Several score systems were created to stratify perioperative risk and predict mortality. The study rises from the needing of a rapid and simple system to identify the patient worthy of Postoperative Intensive Surveillance. In the first phase Authors retrospectively investigated on patients underwent to elective surgery searching for determining factors (DFs) for postoperative ICU admission. Later, Researchers prospectively studied how DFs could predict the admission in ICU of consecutive patients scheduled for elective surgery during a three-months period and created an index, named PoIS (Post-operative Intensive Surveillance), based on the results of this analysis. Authors used surgical invasiveness (SI), Diabetes Mellitus (DM), Myocardiopathy (MCP), Cerebrovascular Disease (CVD), Body Mass Index (BMI), age, serum creatinine level (sCr), Tiffenau Index (TI) and male sex for the development of the original model. Authors classified SI from G1 (lowest) to G5 (highest).

The results show that the power of prediction of postoperative morbidity of PoIS and POSSUM resulted coincident and better than the American Society of Anesthesiology scoring system.

ELIGIBILITY:
Inclusion Criteria:

* elective surgery

Exclusion Criteria:

* multiple surgery
* age less than 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: surgical population
Sampling Method: Non-Probability Sample
Enrollment: 2498 (Actual)
Dates: Start 2015-03; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Post-operative intensive care surveillance scoring system | 1 hour after the end of surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Humanitas Research Hospital - Dept. Anesthesia and Intensive Care Unit, Rozzano, Milano, Italy

IPD SHARING:
Plan to Share IPD: No